CLINICAL TRIAL: NCT01398007
Title: Evaluation of the Efficacy of Camouflage Syringe in Reducing Dental Anxiety and Fear in Children
Brief Title: Use of the Camouflage Syringe to Reduce Dental Anxiety and Fear in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Hospital, India (Other Government)
Collaborators: Lata Medical Research Foundation, Nagpur (Other)
Responsible Party: Principal Investigator, Shweta Ujaoney, Student Dentist, Government Dental College and Hospital, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUT2503
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2011-07

CONDITIONS: Anxiety; Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional syringe (No Intervention): Conventional syringe
- Camouflage syringe (Experimental): The camouflage syringe is divided into three parts: head, body and tail. Head consists of bristles to apply topical anesthesia. The body holds the normally used conventional syringe and presents with a slot to check the aspiration results. The tail hides the conventional syringe loaded with the local anesthetic solution. This syringe is made up of cold-cure acrylic with a colorful toy-like look.
  Interventions: Procedure: Camouflage syringe

INTERVENTIONS:
Procedure: Camouflage syringe — Dental anesthesia is administered using the camouflaged syringe.
  Arms: Camouflage syringe

SUMMARY:
Dental fear and anxiety in children constitue a crucial challenge to dental care delivery as well as future behavior related to dental problems in children. A common cause of such anxiety and fear is the procedural intervention that uses needles and syringes since a visual impact due to the needle acts as a deterrent to the child's cooperation during dental procedures. We therefore improvised the syringe such that it will camouflage the needle. We hypothesized that the use of this needle will alleviate the child's anxiety and therefore will demonstrate improved outcomes related to pain, fear and anxiety. This study is a group randomized trial to test the efficacy of the camouflage syringe as compared to the conventional syringe in children.

DETAILED DESCRIPTION:
The present study was conducted with an aim to evaluate the efficacy of a needle-covering camouflage syringe as compared to the conventional syringe in reducing dental anxiety and fear in children. The study was carried out in 100 children who consecutively reported to the study center and were allocated to the camouflage syringe arm or conventional syringe arm using block randomization to ensure equal distribution across trial arms. The study assessed the degree of dental anxiety and fear using Venham's clinical rating scale in conjunction with rating scale for movement, crying and overall behavior and Venham's Picture Test. The study also assessed parental emotional stress status when the child underwent the injection procedure and the reaction of the child after going home by Parental Emotional Stress Questionnaire and Recall Questionnaire, respectively. The study used appropriate statistical methods to determine the efficacy of the camouflage syringe in reducing the anxiety and fear.

ELIGIBILITY:
Inclusion Criteria:

* Children reporting to study center with dental problems
* Dental procedure requiring local anesthesia
* Informed consent from the parents

Exclusion Criteria:

* Mentally challenged children
* Medical problems negating use of local anesthesia and/or surgical intervention

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2005-10; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Venham's clinical rating scale | Within 1 hour of procedure
  Venham's clinical rating scale for movement, crying and overall behavior

SECONDARY OUTCOMES:
Venham's Picture Test | Within 1 hour of procedure
  Overall aceptability of the intervention
Parental Emotional Stress Questionnaire | Within 1 hour of procedure
Recall questionnaire | Within 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vinay K Hazarey, MDS, Study Chair — Government Dental College and Hospital, India; Jyoti Tote, MDS, Study Director — Government Dental College and Hospital, India; Pushpa V Hazarey, MDS, Study Director — Government Dental College and Hospital, India
Locations (1):
- Government Dental College and Hospital, Nagpur, Maharashtra, India